**Study Protocol** 

Official title of the study: Arteriovenous Fistula Cannulation Practices and Dialysis

Adequacy

NCT number: NCT04270292

Date of document: 20 April, 2020

**Objective:** The aim of this study was to investigate the effect of the cannulation technique

used during needle insertion into the arteriovenous fistula (AVF), the direction of the fistula

needle, the rotation of the needle, the AVF insertion area, and whether the artery and vein

needle are on the same vascular line on the adequacy of the hemodialysis (HD).

**Design:** Descriptive and cross-sectional study

**Methods:** The study was conducted in accordance with the Declaration of Helsinki. The

approval of the local ethics committee approval (Meeting no: 08/042019, Decision no:

P0139R00), permission from the institutions where the study was conducted, and the verbal

consent of the patients were obtained.

This study was conducted between May and December 2019 at the a total of four HD

centers, including one private dialysis center, one private hospital and two state hospitals in

two provinces. The study sample consisted of 164 patients who had received HD treatment

with an AVF for at least six months, at three days a week and four hours a day, were aged 18

years or older, had no problem communicating, and volunteered to participate in the study.

All patients were treated with a high-flux synthetic type dialyzer at the dialysis unit where the

study was conducted. The same dialysate solution was used for each session with a dialysate

temperature of 36°C, a standard bicarbonate concentration 30-35 mmol/l, a dialysate flow rate

500 ml/minute and a pump speed 300-450 ml/minute. All needles placed into the AVF were

of the back eye type. A semi-structured questionnaire form developed by the researchers as a

1

result of a literature survey was used to collect the data. The form included questions on the patients' socio-demographic and clinical data and AVF cannulation. The Kt/V and urea reduction rate (URR) that were used to evaluate dialysis adequacy were regularly evaluated at the HD centers every month and recorded in the patient's chart. The mean three-month Kt /V and URR values starting from the date the study was started were calculated by the researchers and entered into the data form. The questionnaire was then completed by the researchers interviewing the patients with the face-to-face method during the second hour of HD treatment. Completing the forms took about 5 minutes. STROBE check-list was used for reporting the study.

**Statistical Analysis Plan** 

Official title of the study: Arteriovenous Fistula Cannulation Practices and Dialysis

Adequacy

NCT number: NCT04270292

Date of document: 20 April, 2020

**Outcome measures** 

Number of fistula needle direction: The hemodialysis nurse who cannulate the patient's

fistula fill the data form. There is two options about fistula direction as antegrade or

retrograde.

Number of cannulation method: The hemodialysis nurse who cannulate the patient's fistula

fill the data form. There is three options about cannulation method as puncture, buttonhole,

and rope ladder methods.

Number of fistula needle rotated: The researchers look to the fistula needle while it inserts

to the fistula. There is two options as needle rotation is yes or no.

Number of arterial and venous needle been on the same line: The researchers look to the

arterial and venous line whether they are the same venous line.

3

## Results

| Title: | Number of Fistula Needle Direction | | |
|---|---|---|---|
| ▶ Description: | The hemodialysis nurse who cannulate the patient's fistula fill the da | | |
| Time Frame: | e Frame: up to 12 weeks | | |
| ▼ Outcome | ▼ Outcome Measure Data | | |
| ▶ Analysis | Population Descrip | otion | |
| | Arm/Group Title | Arteriovenous Fistula Cannulation Group | |
| ▶ Arm/0 | Group Description: | The cannulation practices' of patie | |
| | Overall Number of ticipants Analyzed | 164 | |
| | easure Type: Count of<br>Participants<br>Measure: participants | | |
| Row Title | | | |
| Α | ntegrade direction | 72 | 43.9% |
| Re | trograde direction | 92 | 56.1% |

| Title: | Number of Cannulation Method | | |
|---|---|---|---|
| ▶ Description: | : The hemodialysis nurse who cannulate the patient's fistula fill the da | | |
| Time Frame: | ime Frame: up to 12 weeks | | |
| ▼ Outcome Measure Data ✓ | | | |
| ▶ Analysis P | ▶ Analysis Population Description | | |
| | Arm/Group Title | Arteriovenous Fistula Cannulation Group | |
| ▶ Arm/Gr | oup Description: | The cannulation practices' of patie | |
| | verall Number of<br>cipants Analyzed | 164 | |
| | asure Type: Count of<br>Participants<br>leasure: participants | | |
| Row Title | | | |
| | Area puncture | 87 | 53.05% |
| | Rope ladder | 54 | 32.93% |
| | Buttunhole | 23 | 14.02% |

| ▼ Outcome Measure Data ▶ Analysis Population Description Arm/Group Title ▶ Arm/Group Description: Overall Number of Participants Analyzed Measure Type: Count of Participants Unit of Measure: participants Row Title Yes Arteriovenous Fistula Cannulation Group 164 Arteriovenous Fistula Cannulation Group 164 164 164 164 164 164 164 16 | | Title: Number of Fistula Needle Rotated Description: The researchers look to the fistula needle while it inserts to the fis Time Frame: up to 12 weeks |
|---|---|---|
| Arm/Group Title Arm/Group Description: Overall Number of Participants Analyzed Measure Type: Count of Participants Unit of Measure: participants Row Title Yes Arteriovenous Fistula Cannulation Group 164 164 164 164 164 164 163.41% | | |
| ► Arm/Group Description: Overall Number of Participants Analyzed Measure: Type: Count of Participants Unit of Measure: participants Row Title Yes The cannulation practices' of patie 164 164 164 164 164 164 164 | ► Analysis Population Descrip | ▶ Analysis Population Description |
| Overall Number of Participants Analyzed Measure Type: Count of Participants Unit of Measure: participants Row Title Yes 104 63.41% | Arm/Group Title | Arteriovenous Fistula Cannulation Group |
| Participants Analyzed Measure Type: Count of Participants Unit of Measure: participants Row Title Yes 104 63.41% | ▶ Arm/Group Description: | The cannulation practices' of patie |
| Participants Unit of Measure: participants Row Title Yes 104 63.41% | | |
| Yes 104 63.41% | Participants | |
| | Yes | 104 63.41% |
| No 60 36.59% | No | 60 36.59% |

| Title: | Number of Arteria | al and Venous Needle Been on the Same Line | |
|---|---|---|---|
| | n: The researchers look to the arterial and venous line whether they are | | |
| Time Frame: | up to 12 weeks | | |
| ▼ Outcome | ▼ Outcome Measure Data ✓ | | |
| ▶ Analysis | Population Descrip | otion | |
| | Arm/Group Title | Arteriovenous Fistula Cannulation Group | |
| ▶ Arm/0 | Group Description: | The cannulation practices' of patie | |
| | Overall Number of ticipants Analyzed | 164 | |
| | easure Type: Count of<br>Participants<br>Measure: participants | | |
| Row Title | | | |
| | Yes | 25 | 15.24% |
| | No | 139 | 84.76% |
| | | | , |

## Statistical analysis

The Statistical Package for Social Sciences (SPSS Inc., Chicago, IL., USA) v. 22.0 software program was used for the statistical analysis of the data from the study. The compliance with a normal distribution of the measurements obtained within the scope of the study was investigated with the "Shapiro-Wilk Test". Mean±standard deviation, median, and interquartile range (IQR) were used to present the descriptive statistics of the continuous numerical variables and number (n) and percentage (%) to present the categorical variables. Values not showing a normal distribution were compared with the "Mann-Whitney U Test" and "Kruskal-Wallis Test", while data with a normal distribution were compared with "Student's t Test" and "One-Way ANOVA". The homogeneity of variances was evaluated with the "Levene test". Pairwise post-hoc comparisons were made by using the "Tukey and Tmahane T2" tests in cases where there was a significant difference between the groups. Independent predictors affecting the Kt/V and URR values were investigated with logistic regression analysis using the possible factors identified with multivariate analysis previously. A p level of 0.05 was accepted as statistically significant in statistical decisions.